CLINICAL TRIAL: NCT07208591
Title: Phase Ⅲ Randomized, Double-blind, Placebo-controlled Evaluation of the Safety and Efficacy of STSA-1002 Injection in Patients With Acute Respiratory Distress Syndrome
Brief Title: To Evaluate The Safety and Efficacy of STSA-1002 Injection in Patients With Acute Respiratory Distress Syndrome
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Staidson (Beijing) Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STSA-1002-07
Record Dates: First submitted 2025-09-28; First posted 2025-10-06 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS)
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients in this group will receive basal treatment and STSA-1002.
  Interventions: Drug: STSA-1002 injection
- Placebo group (Placebo Comparator): Patients in this group will receive basal treatment and STSA-1002.
  Interventions: Drug: STSA-1002 Injection Placebo

INTERVENTIONS:
Drug: STSA-1002 injection — basal treatment + STASA-1002 intravenous infusion
  Arms: Experimental group
Drug: STSA-1002 Injection Placebo — basal treatment + STSA-1002 Injection Placebo
  Arms: Placebo group

SUMMARY:
To evaluate the efficacy, safety and tolerability of STSA-1002 injection in patients with acute respiratory distress syndrome

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old ≤ ≤ 85 years old;
2. laboratory tests results indicate respiratory viral infection;
3. Fulfills the diagnostic criteria for A New Global Definition of Acute Respiratory Distress Syndrome ;
4. The time from the onset of respiratory infection-related symptoms to randomization is ≤ 12 days (for patients without invasive mechanical ventilation)/)/≤ 14 days (for patients with invasive mechanical ventilation); Or worsening of respiratory infection-related symptoms within ≤7 days from randomization;
5. PaO2/FiO2≤200mmHg;
6. The subjects (including their partners) have no plans to have children during the trial and within 3 months after the last dose, and agree to take appropriate and effective contraceptive measures (such as contraceptive pills, condoms, etc.);
7. Volunteer to participate in the trial and sign the informed consent form.

Exclusion Criteria:

1. ECMO before the first dose;
2. According to the comprehensive judgment of the investigator, the patient's condition improved within 48 hours before the first dose;
3. The expected survival period is no more than 24 hours or cardiac arrest occurred 4 weeks before the first dosedose;
4. Patients with stroke or acute coronary syndrome within 3 months before randomization;
5. Patients with cardiogenic pulmonary edema, which is the main cause of respiratory failure; New York Heart Classification III-IV patients;
6. Severe chronic respiratory failure;
7. Known active pulmonary tuberculosis;
8. Combined with liver insufficiency
9. Long-term dialysis and/or known severe renal impairment Cytomegalovirus infection;
10. Known HIV infection with CD4+ T-lymphocyte count < 200 cells/μL;
11. Organ transplant patients;
12. Patients who received radiotherapy and chemotherapy in the past 1 years or the malignant tumor is still in the active phase;
13. Septic shock
14. Absolute neutrophil count is less than 0.5×109/L;
15. Hemoglobin is less than 60g/L, or the researcher judges that there is active gastrointestinal bleeding;
16. Severe underlying diseases with poor compliance with basic treatment;17. Pregnant or lactating women;

18. Participated in new drug clinical trials and medication within 3 months before screening; 19. Allergic or allergic to any component of the trial drug and its excipients (such as allergic to two or more drugs); 20. Other diseases or conditions that the investigator considers unsuitable for participation in this trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
28-day all-cause mortality rate | Day28 after first dose

SECONDARY OUTCOMES:
60-day all-cause mortality rate | Day60 after first dose
Proportion of subjects with a decrease in the level of respiratory support on Day 28 | Day28 after first dose
ICU length of stay and total hospitalization time on Day 28 | Day28 after first dose
Proportion of subjects with PaO2/FiO2 > 300 mmHg or free of respiratory support on Day 28 | Day28 after first dose
Days alive without invasive mechanical ventilation | Day28 after first dose
Changes in SOFA values from baseline on Day 3, 7, 10, and 14 | Day14 after first dose

CONTACTS AND LOCATIONS:
Overall Officials: Bin M.D. Cao, Principal Investigator — China-Japan Friendship Hospital
Locations (15):
- China (15):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Wuhan Central Hospital, Wuhan, Hubei
  - Xiangtan Central Hospital, Xiangtan, Hunan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Weifang People's Hospital, Weifang, Shandong
  - Sichuan Academy of Medical Sciences and Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Dazhou Central Hospital, Dazhou, Sichuan
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang